CLINICAL TRIAL: NCT02555748
Title: Therapeutic Drug Monitoring of Sunitinib and Pazopanib in Advanced or Metastatic Renal Cell Carcinoma
Acronym: SUP-R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14 URO 06
Record Dates: First submitted 2015-09-04; First posted 2015-09-22 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pazopanib (Active Comparator): The daily dose of pazopanib will be the standard dose i.e. 800 mg once a day (2 tablets of 400 mg in one oral administration per day) administered each day, continuously, during the treatment phase (complete cycle will be defined as a 6-week period).
  During the first stage of the study (Part I), adjustment of drug dose will be made according to individual patient tolerance to treatment evaluated by clinical and biological monitoring; During the second stage of the study (Part II), dose modification should also be performed according to individual patient tolerance to treatment evaluated by clinical and biological monitoring ans also by using the new Pharmacokinetic-Pharmacodynamic (PK-PD) Algorithm elaborated during the first part.
  Interventions: Drug: Pazopanib
- Sunitinib (Active Comparator): Sunitinib will be administered at the standard dose of 50 mg, once daily during 4 consecutive weeks, followed by a wash-out period of 2 weeks (corresponding to a complete cycle of 6 weeks).
  During the first stage of the study (Part I), dose adjustment of drug dose will be made according to individual patient tolerance to treatment evaluated by clinical and biological monitoring; During the second stage (Part II), dose modification should also be performed according to individual patient tolerance to treatment evaluated by clinical and biological monitoring ans also by using the new Pharmacokinetic-Pharmacodynamic (PK-PD) Algorithm elaborated during the first part.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Pazopanib
  Arms: Pazopanib
Drug: Sunitinib
  Arms: Sunitinib

SUMMARY:
This pilot study is an open-label interventional study, prospective, non-comparative, sequential (two stages), national, multicenter study.

Patients starting therapy with sunitinib or pazopanib as standard first line treatment for advanced or metastatic renal cell carcinoma will enter the study in one of the two cohorts (115 patients will be treated by sunitinib and 99 patients will be treated by pazopanib).

The purpose of this study is to examine the feasibility of sunitinib and pazopanib dose individualisation based on therapeutic drug monitoring (TDM) and to assess the benefit of this approach in terms of tolerance and efficacy compared with the current empirical method based only on tolerance observation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients starting therapy with sunitinib or pazopanib as standard first line treatment for advanced or metastatic renal cell carcinoma.
2. Measurable tumours as defined by RECIST criteria version 1.1.
3. Age ≥ 18 years old.
4. WHO Performance Status ≤ 2.
5. Life expectancy ≥ 6 months.
6. Adequate cardiac function (baseline Left Ventricular Ejection Fraction (LVEF) ≥ 50% determined by Multiple Gated Acquisition scan (MUGA) or echocardiography) and pulmonary function.
7. Renal function defined as creatinine clearance (Cockcroft and Gault formula) > 30 mL/min.
8. Adequate liver function defined as: total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN); Alanine AminoTansferase (ALAT) and Aspartate AminoTransferase (ASAT) ≤ 2.5 x ULN; Concomitant elevation in bilirubin and ASAT/ALAT above 1.0 x ULN is not allowed.
9. Patients must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up.
10. Negative pregnancy test for women in childbearing potential.
11. Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study (before study entry and until 30 days after the last administration of study treatment).
12. Patients affiliated to a social health insurance.

Exclusion Criteria:

1. Patients without any venous access for blood sampling.
2. Hypersensitivity to the active substance or to any of the excipients.
3. History or clinical evidence of central nervous system (CNS) metastases, except for individuals who have previously-treated CNS metastases.
4. Corrected QT interval (QTc) > 480msecs using Bazett's formula.
5. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, such as, but not limited to:

   * Uncontrolled infection.
   * Cardiovascular conditions within the last 6 months such as cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New-York Heart Association (NYHA), clinically significant irregular heartbeat requiring medication.
   * Poorly controlled hypertension [defined as systolic blood pressure of ≥140 mmHg or diastolic pressure of ≥90 mmHg).
   * History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or deep venous thrombosis (DVT) within the past 6 months.

   Note: patients with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
6. Evidence of active bleeding or bleeding diathesis.
7. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme cytochrome P450 isoenzyme 3A4 (CYP3A4) within the last 14 days prior to inclusion and/or during the study.
8. Patients already treated with an anticancer treatment in the previous four weeks or patient requiring anticancer treatment during the study (chemotherapy, immunotherapy, hormonotherapy, radiotherapy or surgery).
9. Pregnant or breast-feeding women.
10. Positive diagnostic of HIV, B and C hepatitis.
11. Patients with serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with patient's safety, provision of informed consent, or compliance to study procedures.
12. Patients who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Part I: Pharmacokinetics - Pazopanib or Sunitinib plasma concentrations | On day 1 and day 15 during cycle 1 and cycle 2 (cycle length is 6 weeks)
Part II: Tolerance - Proportion of patients without treatment discontinuation due to adverse event (AE) during the first year. | 5.5 years
  This corresponds to the number of patients without treatment discontinuation due to AE among the total number of patients in each group.
Part II: Efficacy - Proportion of patients without progression at 1 year. This corresponds to the number of patients without progression at 1 year among the total number of patients in each group | 5.5 years
Part I: Adverse Events according to NCI toxicity scale (version 4.03) | 1.5 years

SECONDARY OUTCOMES:
Part I and II: Objective Response (e.g. Complete or Partial Response) | 5.5 years
  Objective Response will be defined using RECIST Criteria version 1.1.
Part I and II:- Progression free survival. | 5.5 years
  Progression free survival is defined as the time from inclusion until progression (RECIST Criteria version 1.1) or death. Patients alive at last follow-up news are censored at this date.
Part I and II: Safety according to the classification of the NCI: Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.03. | 5.5 years
Part I and II: Hand-foot syndrome (HFS) | 5.5 years
  Hand-foot syndrome (HFS) will be evaluated using the HFS-14 questionnaire. This scale specifically developed for patients with HFS is a valid and valuable tool for measuring HFS-related QoL impairment.
Part I and II: Quality of life using the quality of life questionnaire (QLQ)-C30 | 5.5 years
  Quality of life will be evaluated using the QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christine CHEVREAU, MD, Principal Investigator — IUCT-O
Locations (8):
- France (8):
  - CHU DE BORDEAUX - Hôpital Saint-André, Bordeaux
  - Institut Bergonie, Bordeaux
  - CHU DE LIMOGES - Hôpital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Regional Du Cancer Montpellier, Montpellier
  - CH RODEZ, Rodez
  - Institut Claudius Regaud, Toulouse